CLINICAL TRIAL: NCT04370210
Title: Sleep Quality During COVID-19 Containment in Children 7 to 12 Years Old, Whether or Not Usually Followed in Child Psychiatry
Brief Title: Sleep Quality During COVID-19 Containment in Children Whether or Not Usually Followed in Child Psychiatry
Acronym: CONFIDODO
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD 0520
Record Dates: First submitted 2020-04-29; First posted 2020-04-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2020-04

CONDITIONS: Sleep Disturbance
Keywords: Children; Sleep Disturbance scale for children; Containment; COVID-19; Anxiety; Psychological Distress; Sleep Wake Disorders; Child Psychiatry; Mental Health
MeSH Terms: conditions — Parasomnias; COVID-19; Anxiety Disorders; Sleep Wake Disorders; Psychological Well-Being | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Child without follow-up in child psychiatry: Child enrolled, and their parents, must complete online questionnaires
  Interventions: Behavioral: Questionnaires
- Child with follow-up in child psychiatry: Child enrolled, and their parents, must complete online questionnaires
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Child of both groups enrolled, and their parents, must complete online questionnaires

SUMMARY:
The purpose of this study is to determine whether sleep disturbances in children aged 7 to 12 during COVID-19 containment are more prevalent in children who received routine psychiatric care before containment compared to children who don't have any psychiatric care.

DETAILED DESCRIPTION:
The coronavirus epidemic reached France in January 2020 and the WHO declared the COVID-19 outbreak was a pandemic on 11 March 2020. In response to this pandemic the French government announced national containment starting on 17 March 2020. Some recent studies suggest that a containment duration of more than 10 days and an extension beyond the originally announced duration would increase the psychological impact of it.

Sleep is a vital function that contributes to the proper neurophysiological and psychological development of human beings especially children. Sleep disorders can have a major impact on a child's behavior, mood, cognitive performance and metabolism. Sleep disorders are often associated with depression, anxiety and cognitive changes. Chronic sleep disorders are also risk factors for mental illness To our knowledge, no study targeting the quality of sleep in children who usually receive psychiatric care is underway or has been published. It is essential to ask what the quality of sleep in children with a psychiatric diagnosis who suddenly lose their bearings and their usual daily routine (school, therapeutic groups, day hospitals, etc.) after several weeks of containment.

This study is designed to assess different parameters in the 2 groups of children (healthy volunteers and Child with follow-up in child psychiatry) :

* the sleep quality,
* the depression level,
* the anxiety level,
* if socio-demographic factors have an influence on sleep disorders,
* if there is a correlation between children's sleep quality, and anxiety level / sleep quality in their parents.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 7 to 11 years and 11 months included on the first day of containment in France on 17 March 2020
* Child receiving care at the CMP of Cergy-le-Haut (medico-psychological center) on the 2020 active patient population (at least one appointment with a child psychiatrist, a psychologist, a psychomotor therapist or a speech therapist or in a therapeutic group between January and March 2020)

OR

* Child not receiving any psychiatric care and having no siblings (half-brother, half-sister) followed in child psychiatry
* No parental opposition

Exclusion Criteria:

* Poor French reading comprehension by parents
* Objection of the child
* Child under guardianship, curatorship or foster care
* Child not on containment : child cared for outside his home everyday (in school and hospital daycare for example).

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Child aged 7 to 11 years and 11 months included on the first day of containment in France on 17 March 2020 and their parents
Sampling Method: Non-Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Comparison of sleep quality during COVID-19 containment between children usually followed in child psychiatry and children without follow-up | An average of 1 day
  Sleep quality is assessed in both groups with the Sleep Disturbance Scale for Children (SDSC scale). A score ≥ 45/125 is considered as pathological.

SECONDARY OUTCOMES:
Assessment of child depression in both groups | An average of 1 day
  Child depression is measured using Child Depression Inventory Scale (CDI scale). For each item the score is graded by severity from 0 (normal behavior) to 2 (severe).
Assessment of child anxiety in both groups | An average of 1 day
  Child anxiety is measured using Revised Children's Manifest Anxiety Scale (RCMAS). For each item, child answer by Yes or No. The total score is interpreted using the correspondence tables in function of sex and age
Assessment of the influence of socio-demographic factors on sleep in both groups | An average of 1 day
  Sleep quality is assessed with the Sleep Disturbance Scale for Children (SDSC scale). The score obtained is interpreted in function of socio-demographic factors (age, sex, lifestyle, couple status, profession and socio-professional category, education)
Measure of the correlation between child sleep quality and parents sleep quality (anxiety level) in both groups | An average of 1 day
  Sleep quality is assessed with the Sleep Disturbance Scale for Children (SDSC scale). For their parents, sleep quality and anxiety level are measured with a numerical scale between 0 and 10. For sleep quality, 0 correspond to a very poor quality and 10 to a very good quality. For anxiety level, 0 correspond to no anxiety and 10 to a severe anxiety. The score obtained for child is interpreted in function of their parents score.
Assessment of sleep disturbance based on psychiatry diagnoses in the group of children usually followed in child psychiatry | An average of 1 day
  Sleep quality is assessed with the Sleep Disturbance Scale for Children (SDSC scale). The score obtained is interpreted in function of child psychiatry diagnoses coded with Diagnostic and Statistical Manual of Mental Disorders (DSM-5)
Assessment of child anxiety based on psychiatry diagnoses in the group of children usually followed in child psychiatry | An average of 1 day
  Child anxiety is measured using Revised Children's Manifest Anxiety Scale (RCMAS). For each item, child answer by Yes or No.
  The score obtained is interpreted in function of child psychiatry diagnoses coded with Diagnostic and Statistical Manual of Mental Disorders (DSM-5)
Assessment of child depression based on psychiatry diagnoses in the group of children usually followed in child psychiatry | An average of 1 day
  Child depression is measured using Child Depression Inventory Scale (CDI scale). For each item the score is graded by severity from 0 (normal behavior) to 2 (severe).
  The score obtained is interpreted in function of child psychiatry diagnoses coded with Diagnostic and Statistical Manual of Mental Disorders (DSM-5)

CONTACTS AND LOCATIONS:
Overall Officials: Erwan VION, Principal Investigator — Hôpital NOVO
Locations (1):
- Centre Hospitalier René Dubos, Pontoise, France

IPD SHARING:
Plan to Share IPD: No